CLINICAL TRIAL: NCT02316535
Title: Low-dose Versus Standard-dose Capecitabine Adjuvant Chemotherapy for Chinese Elderly Patients With Stage II/III Colorectal Cancer: A Randomized, Phase 3 Non-inferiority Study
Brief Title: Low-dose Capecitabine Adjuvant Chemotherapy for Elderly Patients With Stage II/III Colorectal Cancer
Acronym: LcACEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LcACEC-201474
Record Dates: First submitted 2014-12-09; First posted 2014-12-15 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer; stage II/III; elderly; adjuvant chemotherapy; capecitabine; non-inferiority
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard-dose (Active Comparator): capecitabine, oral administration, 1,250 mg/m2 twice daily on days 1-14, and repeated on day 22; 8 circles in total.
  Interventions: Drug: Capecitabine
- reduced-dose (Experimental): capecitabine, oral administration, 1,000 mg/m2 twice daily on days 1-14, and repeated on day 22; 8 circles in total.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — adjuvant chemotherapy;
  Other Names: Xeloda

SUMMARY:
Approximately half of colorectal cancer (CRC) patients were first diagnosed after 70 years old. However, compared with younger patients, elderly patients were often undertreated in chemotherapy due to their impaired tolerance. Recently, there have been great controversy on adjuvant chemotherapy strategy for stage II/III CRC patients. As an oral fluoropyrimidine, capecitabine has been demonstrated to be equivalent to i.v. 5-Fu/leucovorin regimen in stage III CRC patients. In light of fewer adverse effects and better flexibility, capecitabine was regarded as an ideal alternative for elderly CRC patients, but the optimal dosage for stage II/III elderly CRC patients still remains inconclusive. Our trial expected to prospectively randomized 710 postoperative stage II/III elderly CRC patients (between 70 and 90 years of age) to adjuvant mono-chemotherapy with a standard dose of capecitabine (2500 mg/m2/day) or a reduced dose (2000 mg/m2/day). This is a non-inferiority phase 3 trial with a primary endpoint of 3-year disease free survival (DFS), and other outcomes include 3-year overall survival(OS), completion rate, toxic and adverse effects and quality of life(Qol). By this trial, we aimed to achieve more precise evidence on the individualized adjuvant chemotherapy strategy for stage II/III elderly CRC patients.

DETAILED DESCRIPTION:
An estimated 1,200,000 newly diagnosed colorectal cancer(CRC) cases arose worldwide every year, and CRC has become the third most common malignances in China. Especially in urban areas of China, rapid growth of CRC patients has considerably increased the burden of disease. It is well believed that multi-discipline treatment(MDT) including surgery, chemoradiotherapy and target therapy based on individualized characteristics will benefit CRC patients significantly.

Generally, stage II (T3-4N0M0) and stage III (TanyN1-2M0) colorectal carcinoma can be resected by surgery. In 1990s, National Institutes of Health (NIH) suggested that adjuvant chemotherapy should be applied to stage II/III CRC patients to improve their outcomes. As for stage II CRC, results from the QUASA study indicated that adjuvant chemotherapy could improve 5-year overall survival by 3% to 4% for stage II CRC patients. Currently, most of the global guidelines such as National Comprehensive Cancer Network (NCCN) guidelines still recommended adjuvant chemotherapy for stage II/III CRC patients.

In western countries, approximately 50% of the CRC patients were firstly diagnosed after 70 years old. It was reported that in 1980s, the median age of CRC diagnosis in China was 50. However, in 2005 it had reached 58 years old and has kept increasing in recent years. Limited by age-related organ function decline and comorbid conditions, elderly people shows impaired physical and mental tolerance for chemotherapy. Generally for stage II/III CRC patients, both elderly and younger patients shares common principles of chemotherapy, while a large-scale retrospective analysis based on the ACCENT database showed that among all the CRC cases included, patients with the age ≥ 70 only accounted for 17.1%, much lower than normal. Similarly, Shrag and colleagues reported in their investigation that the proportion of patients ≥75 years old undergoing chemotherapy was substantially lower than patients ≤ 75 years old. These evidence implied that elderly CRC patients held much lower acceptance and completion rate of chemotherapy. With respect to outcomes, a pooled analysis including 3351 CRC cases with adjuvant chemotherapy reported no significant difference on both efficacy and adverse effects among groups of various age, indicating elderly patients could achieve the same benefits from adjuvant chemotherapy. Thus, it is essential to improve the acceptance and completion rate by modifying chemotherapy regimen for elderly CRC patients to achieve better prognosis. There was no random controlled trial focusing on the adjuvant chemotherapy for stage II/III elderly CRC patients.

Results of MOSAIC trial showed that adding oxaliplatin to 5-Fu/ leucovorin could significantly improve 5-year survival of stage II/III colon cancer patients, which made the oxaliplatin-based combine chemotherapy (Folfox, Xelox) be recommended by the latest guidelines. In the subgroup analysis of that trial, however, there was no significant improvement detected in stage II patients. Recent analysis from ACCENT database in 2013 indicated that elderly stage II/III CRC patients (≥ 70 yr) acquired no significant benefits from adding oxaliplatin to fluoropyrimidine-based chemotherapy, which suggested monochemotherapy might be a better option for elderly CRC patients.

Capecitabine ( Xeloda®) is the unique oral prodrug of 5-Fu recommended by global guidelines and especially International Society of Geriatric Oncology (SIOG), and it has been verified by clinical trials that in view of efficacy and safety, capecitabine monochemotherapy was equivalent to i.v. 5-Fu/ leucovorin adjuvant chemotherapy. With efficacy retained, a large group of patients prefer capecitabine due to oral administration which can remarkably enhance flexibility and compliance. These advantages make capecitabine a potential ideal choice for elderly patients. According to the NCCN guideline, the standard dosage of capecitabine was 1250mg/m2 .bid. It was well-established that different characteristics such as ethnicity, age and sex could alter the metabolism and change individual tolerance for drugs; hence, there are still controversies on the optimal dose of capecitabine in different populations. The X-Act trial provided a result that among elderly patients (≥ 70 yr) undergoing standard-dose capecitabine adjuvant chemotherapy(1250mg/m2 .bid), 51% of the patients required dose reduction to complete the whole treatment cycle, implying that the recommended 1250mg/m2 .bid. might be an overdose for elderly patients given the fact that only elderly patients with relatively better health (≤ 75 yr, ECOG≤1) were eventually included in X-ACT trial. Chang and colleagues have verified feasibility of a tailored-dose strategy with a starting dose at 1000 mg/m2 .bid in a single-arm study. The European Society for Medical Oncology (ESMO) has also recommended an option of 80% standard dosage (i.e. 1000 mg/m2 .bid) for elderly II/III CRC patients. However, no prospective trial has been conducted yet to confirm this reduced-dose strategy.

Based on current evidence and controversy above, we designed this non-inferiority, phase 3 clinical trial to explore the optimal dosage of capecitabine monochemotherapy for stage II/III elderly CRC patients. Following the results of sample size estimation, 710 postoperative (pT3-4NanyM0 or pTanyN+M0) elderly patients between 70 to 90 years of age were anticipated to be included and randomly divided into two groups (A and B). Patients in group A would receive the standard dose regimen (1,250 mg/m2 twice daily on days 1-14, and repeated on day 22); accordingly the patients in group B would receive the reduced dose regimen (1,000 mg/m2 twice daily on days 1-14, and repeated on day 22). The primary endpoint was 3-year disease free survival (DFS), other outcomes included 3-year overall survival (OS), completion rate, toxic and adverse effects and quality of life (Qol).

ELIGIBILITY:
Inclusion Criteria:

1. With informed consents
2. Histologically identified carcinoma of colon and rectum
3. pT3-4NanyM0 or pTanyN+M0(stage II/III)
4. age between 70 to 90
5. undergone R0 resection
6. ECOG ≤2
7. Stage II patients with microsatellite stable (MSS) or microsatellite low (MSL)

Exclusion Criteria:

1. With other types of malignances simultaneously
2. Creatinine clearance ≤ 70 ml/min
3. Undergone neoadjuvant chemotherapy
4. In anticoagulant therapy
5. Pregnant or lactating women
6. History of antineoplastic drugs
7. With other contraindications for chemotherapy

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
toxic and adverse effects | 30 weeks
completion rate | 24 weeks
quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD/PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Benson AB 3rd, Schrag D, Somerfield MR, Cohen AM, Figueredo AT, Flynn PJ, Krzyzanowska MK, Maroun J, McAllister P, Van Cutsem E, Brouwers M, Charette M, Haller DG. American Society of Clinical Oncology recommendations on adjuvant chemotherapy for stage II colon cancer. J Clin Oncol. 2004 Aug 15;22(16):3408-19. doi: 10.1200/JCO.2004.05.063. Epub 2004 Jun 15. PMID 15199089
- [Background] Quasar Collaborative Group; Gray R, Barnwell J, McConkey C, Hills RK, Williams NS, Kerr DJ. Adjuvant chemotherapy versus observation in patients with colorectal cancer: a randomised study. Lancet. 2007 Dec 15;370(9604):2020-9. doi: 10.1016/S0140-6736(07)61866-2. PMID 18083404
- [Background] Folprecht G, Cunningham D, Ross P, Glimelius B, Di Costanzo F, Wils J, Scheithauer W, Rougier P, Aranda E, Hecker H, Kohne CH. Efficacy of 5-fluorouracil-based chemotherapy in elderly patients with metastatic colorectal cancer: a pooled analysis of clinical trials. Ann Oncol. 2004 Sep;15(9):1330-8. doi: 10.1093/annonc/mdh344. PMID 15319237
- [Background] McCleary NJ, Meyerhardt JA, Green E, Yothers G, de Gramont A, Van Cutsem E, O'Connell M, Twelves CJ, Saltz LB, Haller DG, Sargent DJ. Impact of age on the efficacy of newer adjuvant therapies in patients with stage II/III colon cancer: findings from the ACCENT database. J Clin Oncol. 2013 Jul 10;31(20):2600-6. doi: 10.1200/JCO.2013.49.6638. Epub 2013 Jun 3. PMID 23733765
- [Background] Schrag D, Cramer LD, Bach PB, Begg CB. Age and adjuvant chemotherapy use after surgery for stage III colon cancer. J Natl Cancer Inst. 2001 Jun 6;93(11):850-7. doi: 10.1093/jnci/93.11.850. PMID 11390534
- [Background] Sargent DJ, Goldberg RM, Jacobson SD, Macdonald JS, Labianca R, Haller DG, Shepherd LE, Seitz JF, Francini G. A pooled analysis of adjuvant chemotherapy for resected colon cancer in elderly patients. N Engl J Med. 2001 Oct 11;345(15):1091-7. doi: 10.1056/NEJMoa010957. PMID 11596588
- [Background] Andre T, Boni C, Navarro M, Tabernero J, Hickish T, Topham C, Bonetti A, Clingan P, Bridgewater J, Rivera F, de Gramont A. Improved overall survival with oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment in stage II or III colon cancer in the MOSAIC trial. J Clin Oncol. 2009 Jul 1;27(19):3109-16. doi: 10.1200/JCO.2008.20.6771. Epub 2009 May 18. PMID 19451431
- [Background] Papamichael D, Audisio R, Horiot JC, Glimelius B, Sastre J, Mitry E, Van Cutsem E, Gosney M, Kohne CH, Aapro M; SIOG. Treatment of the elderly colorectal cancer patient: SIOG expert recommendations. Ann Oncol. 2009 Jan;20(1):5-16. doi: 10.1093/annonc/mdn532. Epub 2008 Oct 15. PMID 18922882
- [Background] Van Cutsem E, Hoff PM, Harper P, Bukowski RM, Cunningham D, Dufour P, Graeven U, Lokich J, Madajewicz S, Maroun JA, Marshall JL, Mitchell EP, Perez-Manga G, Rougier P, Schmiegel W, Schoelmerich J, Sobrero A, Schilsky RL. Oral capecitabine vs intravenous 5-fluorouracil and leucovorin: integrated efficacy data and novel analyses from two large, randomised, phase III trials. Br J Cancer. 2004 Mar 22;90(6):1190-7. doi: 10.1038/sj.bjc.6601676. PMID 15026800
- [Background] Hofheinz RD, Wenz F, Post S, Matzdorff A, Laechelt S, Hartmann JT, Muller L, Link H, Moehler M, Kettner E, Fritz E, Hieber U, Lindemann HW, Grunewald M, Kremers S, Constantin C, Hipp M, Hartung G, Gencer D, Kienle P, Burkholder I, Hochhaus A. Chemoradiotherapy with capecitabine versus fluorouracil for locally advanced rectal cancer: a randomised, multicentre, non-inferiority, phase 3 trial. Lancet Oncol. 2012 Jun;13(6):579-88. doi: 10.1016/S1470-2045(12)70116-X. Epub 2012 Apr 13. PMID 22503032
- [Background] Twelves C, Wong A, Nowacki MP, Abt M, Burris H 3rd, Carrato A, Cassidy J, Cervantes A, Fagerberg J, Georgoulias V, Husseini F, Jodrell D, Koralewski P, Kroning H, Maroun J, Marschner N, McKendrick J, Pawlicki M, Rosso R, Schuller J, Seitz JF, Stabuc B, Tujakowski J, Van Hazel G, Zaluski J, Scheithauer W. Capecitabine as adjuvant treatment for stage III colon cancer. N Engl J Med. 2005 Jun 30;352(26):2696-704. doi: 10.1056/NEJMoa043116. PMID 15987918
- [Background] Chang HJ, Lee KW, Kim JH, Bang SM, Kim YJ, Kim DW, Kang SB, Lee JS. Adjuvant capecitabine chemotherapy using a tailored-dose strategy in elderly patients with colon cancer. Ann Oncol. 2012 Apr;23(4):911-8. doi: 10.1093/annonc/mdr329. Epub 2011 Aug 4. PMID 21821549
- [Derived] He Y, Liu P, Zhang Y, Deng X, Meng W, Wei M, Yang T, Wang Z, Qiu M. Low-dose capecitabine adjuvant chemotherapy in elderly stage II/III colorectal cancer patients (LC-ACEC): study protocol for a randomized controlled trial. Trials. 2015 May 29;16:238. doi: 10.1186/s13063-015-0753-7. PMID 26021722